CLINICAL TRIAL: NCT06691932
Title: At-the-Breast vs. Expressed Human Milk: Genesis of Infant Nutrition (BEGIN)
Acronym: BEGIN
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Bridget Young, Associate Professor of Pediatrics, University of Rochester
Other Study IDs: STUDY00007528; R01HD112363 (NIH)
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Breast Feeding; Exclusive Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers primarily feeding their baby expressed HM (Express Group)
- Mothers primarily feeding their baby directly at-the-breast (ATB Group)

SUMMARY:
The purpose of this study is to define human milk (HM) as an ecosystem which investigators will then combine into temporal models of milk dynamics to accurately describe HM chronobiology. This study addresses 4 crucial public health gaps: 1) how breast milk changes over time and over the day, 2) how milk dynamics are related to infant sleep patterns, 3) how milk dynamics are related to infant microbiome dynamics, and 4) how all these relationships differ between infants fed directly at-the-breast vs pumped milk. These fundamental insights have been unknown until now, so that families who feed pumped breast milk are completely underserved. These results are critical to optimizing infant feeding and health outcomes for all infants receiving breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Lactating mothers between 20-40 years old at enrollment

  o 120 mother/infant dyads who primarily feed HM ATB (average >75% of feeds,
* pumping no more than one time per day)

  o 120 mother/infant dyads who predominantly feed expressed HM (average >75% of feeds)
* All races and ethnicities may enroll
* Singleton infant delivered after 37 weeks
* Infant between the ages of 0-1 months at the time of enrollment.
* No serious health complications in mother or infant

Exclusion Criteria:

* Non-English-speaking subjects as study personnel only speak English
* Lactating moms who will be feeding both ATB and expressed HM (over 25% of the time in either feeding mode)
* Infant supplementation with formula ≥10 oz before sample collections begin, and/or no more than 16 oz during active participation/ sample collections.

Ages: 0 Days to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: 240 mother/infant dyads exclusively feeding HM to healthy infants between 1-5 months postpartum: 120 mothers primarily feeding ATB (ATB Group) and 120 mothers predominantly feeding expressed HM (Express Group)
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Infant Sleep Latency | Baseline, 2 months and 4 months
  The time to fall asleep after bedtime(minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States